CLINICAL TRIAL: NCT01302964
Title: Mirtazapine Treatment of Anxiety in Children and Adolescents With Pervasive Developmental Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Christopher John McDougle, M.D., Director, Lurie Center for Autism, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P001009
Record Dates: First submitted 2010-08-25; First posted 2011-02-24 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Autism Spectrum Disorders
Keywords: Autistic Disorder; Asperger's Disorder; Pervasive Developmental Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive | interventions — Sugars; Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirtazapine (Experimental): The starting dose for subjects is 7.5 mg daily. The maximum daily dose will be 45 mg.
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): Subjects randomized to placebo arm will receive capsules identical in size and appearance to those subjects receiving study drug. Placebo capsules contain inactive ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Subjects randomized to placebo will receive placebo for duration of the study
  Other Names: Sugar pill
  Arms: Placebo
Drug: Mirtazapine — Subjects will receive 7.5 mg daily at the start of the trial. The dose will be increased by 7.5 mg per week for subjects weighing less than 50 kg and up to 15 mg per week for subjects weighing more than 50 kg depending on efficacy and tolerability.
  Other Names: Remeron
  Arms: Mirtazapine

SUMMARY:
This study will determine the effectiveness of mirtazapine in reducing anxiety in children with autistic disorder, Asperger's disorder and Pervasive Developmental Disorder.

DETAILED DESCRIPTION:
One of the areas receiving very little attention in Pervasive Developmental Disorders (PDDs) is that of anxiety. Anxiety is common in PDD, but has not yet been fully characterized. The primary objective of this study is to conduct a preliminary placebo-controlled trial of mirtazapine for the treatment of anxiety associated with PDDs. We hypothesize that mirtazapine will be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-17 years
* Diagnosis of autistic disorder, Asperger's disorder or Pervasive Developmental Disorder Not Otherwise Specified (PDD NOS)
* Clinically significant anxiety as evidenced by a Pediatric Anxiety Rating Scale (PARS) score of 10 or greater
* Abbreviated intelligence quotient (IQ) greater than 50 on the Stanford Binet 5th Ed.

Exclusion Criteria:

* Diagnosis of Rett's disorder or childhood integrative disorder
* Diagnosis of obsessive-compulsive disorder (OCD), post-traumatic stress disorder, major mood disorder, psychotic disorder, or substance use disorder
* Presence of any past or present medical conditions that would make treatment with mirtazapine unsafe
* Use of other antidepressants or benzodiazepines
* Use of other psychotropic medications which are ineffective, poorly tolerated, or sub-optimal in terms of dose
* Previous adequate trial of mirtazapine

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. McDougle, M.D., Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Riley Child and Adolescent Psychiatry Clinic Riley Hospital, Indianapolis, Indiana
  - Lurie Center -MassGeneral Hospital, Lexington, Massachusetts

REFERENCES:
- [Derived] McDougle CJ, Thom RP, Ravichandran CT, Palumbo ML, Politte LC, Mullett JE, Keary CJ, Erickson CA, Stigler KA, Mathieu-Frasier L, Posey DJ. A randomized double-blind, placebo-controlled pilot trial of mirtazapine for anxiety in children and adolescents with autism spectrum disorder. Neuropsychopharmacology. 2022 May;47(6):1263-1270. doi: 10.1038/s41386-022-01295-4. Epub 2022 Mar 3. PMID 35241779

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirtazapine: The starting dose for subjects is 7.5 mg daily. The maximum daily dose will be 45 mg.
  Mirtazapine: Subjects will receive 7.5 mg daily at the start of the trial. The dose will be increased by 7.5 mg weekly for subjects weighing less than 50 kg and up to 15 mg weekly for subjects weighing more than 50 kg depending upon efficacy and tolerability.
Period: Overall Study
Arm/Group | Mirtazapine | Placebo
Started | 20 | 10
Completed | 19 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirtazapine | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (3.6) | 11.3 (4.1) | 11.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 17 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 16 | 8 | 24
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 9 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean 10-Week Change in Pediatric Anxiety Rating Scale 5-Item Total Score, Double-blind Phase
Description: The Pediatric Anxiety Rating Scale (PARS) is a clinician-rated instrument that assesses anxiety symptoms that are commonly associated with social anxiety, separation anxiety, and generalized anxiety disorders. Scaled score ranges form 0-25 with higher scores indicating more severe anxiety symptoms. Means were estimated using a repeated measures linear regression model with treatment group, study week (in categories), and their interaction as covariates, and assuming a common mean between treatment groups at baseline. Confidence intervals reflect a Bonferroni multiple testing correction accounting for the selection of two primary outcomes.
Time Frame: Weeks Baseline, 2, 4, 6, and 10
Population: All randomized study participants
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Mirtazapine: The starting dose for subjects is 7.5 mg daily. The maximum daily dose will be 45 mg.
  Mirtazapine: Subjects will receive 7.5 mg daily at the start of the trial. The dose will be increased by 7.5 mg weekly for subject weighing less than 50kg and up to 15 mg weekly for subjects weighing more than 50kg depending upon efficacy and tolerability.
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale | -4.9 [-7.3 to -2.6] | -3.2 [-6.5 to 0.2]

2. Primary Outcome: Proportion of Participants Who Responded to Treatment at 10 Weeks According to the Improvement Item of the Clinical Global Impression-Scale (Response Defined as CGI-I=1 or CGI-I=2)
Description: The Clinical Global Impressions Global Improvement (CGI-I) is designed to take into account all factors to arrive at an assessment of response to treatment. The CGI-I scale ranges from 1 to 7 (1=very much improved; 2= much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse), with lower scores indicating improvement (1=very much improved and 2=much improved). In this study the CGI was focused on the target symptom of anxiety. Participants with a CGI-I score of 1 or 2 were classified as responders. The CGI-I was administered biweekly for 6 weeks and again at 10 weeks during the study. The participant who withdrew from the study before 10 weeks was not included in the calculations.
Time Frame: Screen (Visit 1) Baseline (Visit 2) and Endpoint (Week 10)
Population: All randomized study participants with a 10 week CGI-I rating
Measure: Number; unit: Proportion of participants
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 19 | 10
Proportion of participants | 0.47 | 0.20

ADVERSE EVENTS:
Time Frame: Ten weeks or at the time of latest data collection for the participant who did not complete the study.
Description: Adverse event information was collected via a structured side effect rating scale completed with the participant and their primary caregiver. This included a list of side-effects that have been reported with mirtazapine at a rate greater than 1%. The physician also asked about any visits to the doctor, new medication use, or any other complaints. Events that were not present at baseline and occurred or worsened after the date of randomization are reported.
Arm/Group | Mirtazapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 20/20 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mirtazapine (N=20) | Placebo (N=10)
Eye Irritation (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 3
Diarrhea (Gastrointestinal disorders) | 5 | 2
Stomach or abdominal discomfort (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 3 | 3
Taste abnormality (Gastrointestinal disorders) | 1 | 0
Indigestion (Gastrointestinal disorders) | 0 | 1
Sedation/Drowsiness (General disorders) | 12 | 6
Appetite increase (General disorders) | 10 | 2
Appetite decrease (General disorders) | 2 | 2
Fever (General disorders) | 2 | 2
Dry mouth (General disorders) | 2 | 0
Tiredness/fatigue (General disorders) | 2 | 0
Accidental injury (General disorders) | 1 | 0
Other Pain (General disorders) | 1 | 0
Allergies Not Otherwise Specified (Immune system disorders) | 1 | 1
Nasal congestion or Cold (Infections and infestations) | 4 | 2
Unspecified or not otherwise listed nose/throat (Infections and infestations) | 2 | 1
Sinus condition (Infections and infestations) | 2 | 0
Flu or upper respiratory problems (Infections and infestations) | 0 | 2
Ear Infection (Infections and infestations) | 1 | 0
Sore throat (Infections and infestations) | 1 | 0
Throat infection (Infections and infestations) | 1 | 0
Unspecified or not otherwise listed mouth (Infections and infestations) | 0 | 1
Unspecified or not otherwise listed, musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Sensory sensitivity (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 5 | 4 — Aggression (e.g. verbal threats to harm others, physical aggressions, not including disobedience or defiant/oppositional behavior)
Nightmares or Dreams (Psychiatric disorders) | 4 | 2
Irritability (Psychiatric disorders) | 7 | 3
Sadness (Psychiatric disorders) | 4 | 3
Difficulty falling asleep (Psychiatric disorders) | 3 | 1
Interrupted sleep/other sleep problems (Psychiatric disorders) | 2 | 0
Concentration difficulty (Psychiatric disorders) | 2 | 1
Anxiety/Nervousness/Worry (Psychiatric disorders) | 2 | 0
Body-focused repetitive behavior (Psychiatric disorders) | 2 | 0
Change in speech (Psychiatric disorders) | 2 | 0
Euphoria/Giddiness (Psychiatric disorders) | 1 | 0
Increased motor activity (Psychiatric disorders) | 1 | 0
Restlessness/Agitation including fidgety (Psychiatric disorders) | 1 | 1
Unspecified or not otherwise listed psych (Psychiatric disorders) | 1 | 0
Decreased motor activity (Psychiatric disorders) | 1 | 0
Suicidal ideas (Psychiatric disorders) | 1 | 0
Social withdrawal (Psychiatric disorders) | 2 | 2
Stereotypy (Psychiatric disorders) | 1 | 1
Enuresis (Renal and urinary disorders) | 3 | 1
Localized rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hair problems (Skin and subcutaneous tissue disorders) | 1 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
Dizziness/faintness (Vascular disorders) | 2 | 1
Intermittent nosebleed (Vascular disorders) | 1 | 0
Compulsions (Psychiatric disorders) | 1 | 0
Disinhibition (Psychiatric disorders) | 1 | 0
Emotional outburst (Psychiatric disorders) | 1 | 0
Self-injurious behavior (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT01302964/Prot_SAP_000.pdf